CLINICAL TRIAL: NCT04171739
Title: A Phase I, Open Label Study in Healthy Subjects to Evaluate the Effect of Itraconazole and Rifampicin Upon the Pharmacokinetics of a Single Oral Dose of Olorofim.
Brief Title: Drug-drug Interaction (DDI) Study to Assess Effect of Itraconazole and Rifampicin Upon Olorofim
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F901318-01-15
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2019-11

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole; Rifampin; olorofim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Other): Itraconazole DDI
  Interventions: Drug: Itraconazole oral solution; Drug: Olorofim
- Cohort B (Other): Rifampicin DDI
  Interventions: Drug: Rifampicin Oral Capsule; Drug: Olorofim

INTERVENTIONS:
Drug: Itraconazole oral solution — 200 mg once daily on Days 6 to 15
  Arms: Cohort A
Drug: Rifampicin Oral Capsule — 600 mg once daily on Days 6 to 15
  Arms: Cohort B
Drug: Olorofim — Single oral dose on Days 1 and 11
  Other Names: F901318

SUMMARY:
This is a Phase 1, single-centre, fixed-sequence, open label, drug-drug interaction study in 2 groups of healthy subjects.

Group A: to evaluate the effects of itraconazole, a strong inhibitor of cytochrome P450 3A (CYP3A), upon the pharmacokinetics of olorofim .

Group B: t o evaluate the effects rifampicin, a strong inducer of CYP3A, upon the pharmacokinetics of olorofim .

ELIGIBILITY:
Inclusion Criteria:

* males or females of any ethnic origin between 18 and 55 years of age
* subjects weighing between 50 and 100 kg, with a body mass index (BMI) between 18 and 32 kg/m2.
* subjects in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations

Exclusion Criteria:

* Female subjects of child-bearing potential.
* Male subjects (or their partners) who are not willing to use appropriate contraception during the study and for 3 months after end of dosing.
* Female subjects who are pregnant or lactating.
* Subjects who have received any prescribed systemic or topical medication within 14 days of first dose administration
* Subjects who have used any non-prescribed systemic or topical medication within 7 days of first dose administration
* Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of first dose administration
* Subjects with or history of clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatry, respiratory, metabolic, endocrine, ocular haematological or other major disorders as determined by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration (Cmax) for olorofim. | 16 days
Area under the concentration-time curve to time of last quantifiable concentration (AUC0-tlast) for olorofim. | 16 days

SECONDARY OUTCOMES:
Time to Cmax (Tmax) of olorofim | 16 days
area under the concentration-time curve to infinity (AUC0-∞) for olorofim | 16 days
terminal elimination half-life (t½) for olorofim | 16 days
Number of subjects with treatment-related adverse events | 23 days

CONTACTS AND LOCATIONS:
Overall Officials: Adeep Puri, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No